CLINICAL TRIAL: NCT00429065
Title: Selection of Young Patients (< 61 Years), With Good Prognosis Diffuse Large B Cell Lymphoma, According to the Immunophenotype (BCL-6 Negative) to be Treated With Chemoimmunotherapy, With R-CHOP. A Pilot Study.
Brief Title: Treatment of Good Prognosis, BCL-6 Negative Diffuse Large Cell Lymphoma With CHOP-R in Patients < 61 Years Old.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Other Study IDs: Hemato INCAN 01/2007
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2007-01-31 (Estimated); Status verified 2007-01

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Non-Hodgkin lymphoma; rituximab; immunotherapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
The purpose of this study is to determine whether a specific subtype of lymphoma responds optimally to treatment with rituximab and chemotherapy.

DETAILED DESCRIPTION:
Treatment with rituximab and chemotherapy (R-CHOP)is the accepted treatment for young patients with diffuse large B cell Non-Hodgkin's Lymphoma. However not every patient benefits with this expensive therapy. Recent data suggest that patients with BCL-6 negative lymphoma are more sensitive to Rituximab therapy. It is also known that patients with high-intermediate and high IPI risk does not benefit form standard three weekly CHOP chemotherapy.

In this study we intend to define a subgroup of patients in whom this therapy will be of maximum benefit.

We will prospectively treat a group of patients with the following characteristics:

< 60 years old low and low intermediate IPI risk BCL-6 negative B-cell NHL Treatment regimen: R-CHOP (standard dosis) for 8 cycles

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Large B cell Non-Hodgkin Lymphoma CD20+
* BCL-6 negative
* Age < 61 years old
* ECOG 2 or less
* IPI low, low intermediate
* Stage II, III or IV
* Signed Informed Consent

Exclusion Criteria:

* Stage I
* Previous treatment
* Lymphomatous central nervous system involvement
* Heart disease
* Kidney failure (serum creatinine > 2 mg/dl)
* HIV +
* Viral Hepatitis
* Pregnancy

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2007-01; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Sobrevilla-Calvo, MD, Principal Investigator — Instituto Nacional de Cancerologia Mexico; Silvia Rivas-Vera, MD, Principal Investigator — Instituto Nacional de Cancerologia Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, D.F., Mexico

REFERENCES:
- [Background] Winter JN, Weller EA, Horning SJ, Krajewska M, Variakojis D, Habermann TM, Fisher RI, Kurtin PJ, Macon WR, Chhanabhai M, Felgar RE, Hsi ED, Medeiros LJ, Weick JK, Reed JC, Gascoyne RD. Prognostic significance of Bcl-6 protein expression in DLBCL treated with CHOP or R-CHOP: a prospective correlative study. Blood. 2006 Jun 1;107(11):4207-13. doi: 10.1182/blood-2005-10-4222. Epub 2006 Jan 31. PMID 16449523
- [Background] Lossos IS, Jones CD, Warnke R, Natkunam Y, Kaizer H, Zehnder JL, Tibshirani R, Levy R. Expression of a single gene, BCL-6, strongly predicts survival in patients with diffuse large B-cell lymphoma. Blood. 2001 Aug 15;98(4):945-51. doi: 10.1182/blood.v98.4.945. PMID 11493437
- [Background] Lossos IS, Czerwinski DK, Alizadeh AA, Wechser MA, Tibshirani R, Botstein D, Levy R. Prediction of survival in diffuse large-B-cell lymphoma based on the expression of six genes. N Engl J Med. 2004 Apr 29;350(18):1828-37. doi: 10.1056/NEJMoa032520. PMID 15115829